CLINICAL TRIAL: NCT05661201
Title: Phase I Study of NEROFE and Doxorubicin in KRAS-mutated ST2-positive Solid Tumors
Brief Title: NEROFE and Doxorubicin in KRAS-mutated ST2-positive Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Immune System Key Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005711
Record Dates: First submitted 2022-11-28; First posted 2022-12-22 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor; KRAS Mutation-Related Tumors
MeSH Terms: interventions — tumor-cells apoptosis factor, human; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Level 1: NEROFE with doxorubicin (Experimental): weekly doses of NEROFE at 96 mg/m2, intravenously over 60 minutes
  Interventions: Drug: NEROFE; Drug: Doxorubicin
- Dose level -1: Nerofe with doxorubicin (Experimental): weekly doses of NEROFE at 48 mg/m2, intravenously over 60 minutes
  Interventions: Drug: NEROFE; Drug: Doxorubicin
- Dose level 2: Nerofe with doxorubicin (Experimental): weekly doses of NEROFE at 192 mg/m2, intravenously over 60 minutes
  Interventions: Drug: NEROFE; Drug: Doxorubicin
- Dose Level 3: Nerofe with doxorubicin (Experimental): weekly doses of NEROFE at 288 mg/m2, intravenously over 120 minutes
  Interventions: Drug: NEROFE; Drug: Doxorubicin
- Dose Level 4: Nerofe with doxorubicin (Experimental): twice weekly doses of NEROFE at 288 mg/m2, intravenously over 120 minutes
  Interventions: Drug: NEROFE; Drug: Doxorubicin

INTERVENTIONS:
Drug: NEROFE — weekly doses of NEROFE (48-288 mg/m2) (dose level 1: 96 mg/m2, dose level -1: 48 mg/m2, dose level 2: 192 mg/m2, dose level 3: 288 mg/m2), intravenously over 60 minutes
Drug: Doxorubicin — weekly doses of 8 mg/m2 (fixed dose), intravenous push over 3 mins;
  Other Names: adriamycin

SUMMARY:
The goal of this clinical trial is to learn about the safety of NEROFE and doxorubicin and how well it works in patients with advanced/unresectable or metastatic solid KRAS-mutated and ST-positive solid tumors. The main question it aims to answer is to find the recommended dose and scheduled for the combination of NEROFE and doxorubicin. Participants will receive weekly doses of NEROFE and doxorubicin.

ELIGIBILITY:
Inclusion Criteria:

* Advanced/unresectable or metastatic solid tumor with a pathogenic KRAS mutation via polymerase chain reaction (PCR), next-generation sequencing (NGS), or other standard test (blood-based DNA testing is allowed)
* Presence of tumor ST2 expression via immunochemistry assay
* Progression or intolerance to all standard therapies, patient may decline standard therapies and retain eligibility (patients must not have available curative options); patients must have been exposed to 2 or fewer lines of systemic therapy for advanced disease (these patients would decline any unused standard therapies which are still available)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Laboratory inclusion criteria:

  * Absolute neutrophil count ≥ 1500/mm3
  * Hemoglobin ≥ 9.0 g/dL (transfusions are allowed to achieve this inclusion criterion)
  * Platelets ≥ 100 x 109/L (transfusions are NOT allowed to achieve this inclusion criterion)
  * Creatinine clearance ≥ 50 mL/min/1.73 m2 using the formula: creatinine clearance = [[140 - age(yr)]*weight(kg)]/[72*serum Cr(mg/dL)] (multiply by 0.85 for women).
  * AST and ALT ≤ 3 x the upper limit of normal of the institution's normal range and total bilirubin ≤ 1.5 x the upper limit of normal of the institution's normal range - if liver metastases are present, AST and ALT ≤ 5 x the upper limit of normal of the institution's normal range and total bilirubin ≤ 3 x the upper limit of normal of the institution's normal range unless there is persistent nausea, vomiting, right upper quadrant pain, fever, rash, or eosinophilia
  * Partial Thromboplastin Time (PTT) must be ≤ 1.5 × upper limit of normal of institution's normal range and INR (International Normalized Ratio) < 1.5. Subjects on anticoagulation (such as warfarin) will be permitted to enroll as long as the INR is in the acceptable therapeutic range as determined by the investigator
* Patients must have fully recovered from all effects of surgery. Patients must have had at least two weeks after minor surgery and four weeks after major surgery before starting therapy. Minor procedures requiring "twilight" sedation such as endoscopies or mediport placement may only require a 24-hour waiting period, but this must be discussed with an investigator
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment and/or postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
* Patient is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by the Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures
* Have measurable disease by RECIST v. 1.1
* Have disease amenable to serial core tumor biopsies
* Suitable, stable venous access to allow for all study-related blood sampling (a central line such as a portacath (e.g. Medi-Port) or PICC is highly encouraged)

Exclusion Criteria:

* Age < 18 years
* Prior exposure to anthracycline chemotherapy
* Receiving any active anti-cancer therapy while on study treatment
* Brain metastases unless they have been previously treated with surgery and/or radiation at least 4 weeks prior to C1D1 and have a baseline MRI that shows no evidence of active/progressing intracranial disease
* Anti-tumor therapy within 3 weeks of C1D1 (defined as, but not limited to, cytotoxic chemotherapy, immunotherapy, biological therapy, radiotherapy, and investigational agents), the "wash-out period"
* Concurrent severe illness or uncontrolled medical condition that, in the investigator's judgement, would cause unacceptable safety risks
* Women who are pregnant or breastfeeding
* Concurrent use of an aromatase inhibitor
* Psychiatric illness or social situation that would limit compliance with study requirements
* Concurrent malignancy or malignancy within 2 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer, or a malignancy that the investigator deems has been definitively treated (e.g. early stage prostate cancer)
* Active hepatitis B, C, or HIV (patients with hepatitis C infection are eligible if they have an undetectable viral load following definitive treatment, patients with HIV are eligible if they have an undetectable viral load and a CD4 count above 500 cells/mm3)
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
  * Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
  * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block)
  * QTcF (using Fridericia's correction) of > 480 msec
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

    1. Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
    2. Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication
    3. Inability to determine the QT interval on screening (QTcF, using Fridericia's correction)
  * Systolic blood pressure (SBP) >160 mmHg or <90 mmHg at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Cycle 1 Day 1 until 30 days following discontinuation of study drug, approximately 6 months.
  Safety and tolerability of NEROFE and doxorubicin in patients with advanced KRAS-mutated and ST2-positive solid tumors
Incidence of Serious Adverse events | From time of Consent until 30 days following discontinuation of study drug, approximately 6 months.
  Safety and tolerability of NEROFE and doxorubicin in patients with advanced KRAS-mutated and ST2-positive solid tumors
Incidence of Adverse events meeting protocol defined dose limiting toxicities | Cyce 1 Day 1 through 28 days
  Safety and tolerability of NEROFE and doxorubicin in patients with advanced KRAS-mutated and ST2-positive solid tumors

SECONDARY OUTCOMES:
Pharmacokinetic (PK): AUC (area under the curve) 0-24 hours | 24 hours, on Cycle 1 Day 1 and Cycle 2 Day 1 (each cycle is 28 days)
  Pharmacokinetics of NEROFE and doxorubicin in patients with advanced KRAS-mutated and ST2-positive solid tumors; AUC 0-24 hours calculated using the trapezoidal rule [(Concentration at 0 hour + concentration at 24 hours) x 24]/2
Pharmacokinetic: Cmax | 24 hours, on Cycle 1 Day 1 and Cycle 2 Day 1 (each cycle is 28 days)
  Pharmacokinetics of NEROFE and doxorubicin in patients with advanced KRAS-mutated and ST2-positive solid tumors; maximum 24 hour concentration
Pharmacokinetic: Cmin | 24 hours, on Cycle 1 Day 1 and Cycle 2 Day 1 (each cycle is 28 days)
  Pharmacokinetics of NEROFE and doxorubicin in patients with advanced KRAS-mutated and ST2-positive solid tumors; minimum 24 hours concentration
Pharmacokinetic: Tmax | 24 hours, on Cycle 1 Day 1 and Cycle 2 Day 1 (each cycle is 28 days)
  Pharmacokinetics of NEROFE and doxorubicin in patients with advanced KRAS-mutated and ST2-positive solid tumors; hour at which Cmax occurs
Pharmacokinetic: t1/2 | 24 hours, on Cycle 1 Day 1 and Cycle 2 Day 1 (each cycle is 28 days)
  Pharmacokinetics of NEROFE and doxorubicin in patients with advanced KRAS-mutated and ST2-positive solid tumors; the time at which the concentration is at half its initial value
Pharmacodynamics: Change in ST2 expression | pretreatment to Cycle 2 Day 15 (each cycle is 28 days)
  Pharmacodynamics of NEROFE and doxorubicin in patients with advanced KRAS--mutated and ST2-positive solid tumors; Change in ST2 expression by IHC will be quantified by percentage of positively stained cells in pre- vs. on-treatment tumor biopsies
Pharmacodynamics: Change in KRAS mRNA | pretreatment to Cycle 2 Day 15 (each cycle is 28 days)
  Pharmacodynamics of NEROFE and doxorubicin in patients with advanced KRAS-mutated and ST2-positive solid tumors; Change in KRAS mRNA will be quantified by qPCR in blood and tissue (pre- vs. on-treatment blood samples and tumor biopsies).
Progression free survival (PFS) | 6 months
  time from the date of the initial treatment to the date of first documented disease progression or death due to any cause, whichever occurs first.
Overall Survival (OS) | 2 years 6 months
  Overall Survival (OS): defined as the date of the initial treatment to the date of the participant's death.
Overall Response Rate (ORR) | every 8 weeks until progression, approximately 6 months
  The proportion of participants who achieve a PR or better according to the RECIST version 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Weinberg, MD, Study Chair — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No